CLINICAL TRIAL: NCT05403099
Title: Effect of Topical Application of Hyaluronic Acid on Stability of Immediate Loading Dental Implant in Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 01010119
Record Dates: First submitted 2022-05-20; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Missing Teeth
Keywords: Hyaluronic Acid, dental implant
MeSH Terms: conditions — Anodontia | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Twenty implants were inserted in patients seeking for replacement of missed single or multiple posterior maxillary teeth. Patients were divided randomly into two groups. In the control group, ten implants were placed and immediately loaded. While in the study group, ten implants were coated with hyaluronic acid (HA) immediately before placement and immediately loaded. All patients were clinically evaluated at implant placement time, one, three and six months after loading regarding implant stability. Peri-implant pocket depth and modified sulcus bleeding index were evaluated clinically at six months in all patients. Bone density was evaluated radiographically after three months. All clinical and radiographic data were subjected to statistical analysis.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Each implant was placed into the prepared implant site.
  Interventions: Other: conventional implant placement
- Hyaluronic acid (Experimental): Each implant was placed after topical application of HA on its surface
  Interventions: Other: Hyaluronic acid

INTERVENTIONS:
Other: Hyaluronic acid — immediate placement of dental implant after topical application of hyaluronic acid on implant surface
  Arms: Hyaluronic acid
Other: conventional implant placement — immediate placement of dental implant without application of hyaluronic acid on implant surface
  Arms: control

SUMMARY:
Effect of Topical Application of Hyaluronic Acid on Stability of Immediate Loading Dental Implant in Posterior Maxilla

DETAILED DESCRIPTION:
Patients were randomly divided into two groups:

Group I (Control group):

Ten implants were placed in posterior maxilla and immediately loaded.

Group II (Study group):

Ten implants were coated with HA before placement in posterior maxilla and immediately loaded.

ELIGIBILITY:
Inclusion Criteria:

* Highly motivated patients with good oral hygiene.
* Age 18 years or older.
* Adequate alveolar bone volume at the implant site, at least 6mm in width and 15 mm in height.
* Free from any parafunctional habits

Exclusion Criteria:

* Patients suffering from any systemic or local disease that contraindicate implant placement or surgery.
* Pregnancy.
* Smokers.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
implant stability | immediately after surgery
  using radiofrequency analysis
implant stability | one month
  using radiofrequency analysis
implant stability | three months
  using radiofrequency analysis
implant stability | six months
  using radiofrequency analysis
bone density | three months
  bone density around the implant is measured in cone beam computed tomography

SECONDARY OUTCOMES:
propping depth | six months
  The distance between the gingival margin and the base of the pocket
bleeding inex | six months
  Modified sulcus bleeding index

CONTACTS AND LOCATIONS:
Locations (1):
- Merna Elhadidi, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No